CLINICAL TRIAL: NCT03411499
Title: Stroke-free Survival Comparison Between Early Surgery and Conventional Therapy in Left Infective Endocarditis - A Multicenter Partially Randomized Preference Trial (EARLY Study)
Brief Title: Stroke-free Survival Comparison Between Early Surgery and Conventional Therapy in Left Infective Endocarditis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped because of low enrollment.
Sponsor: Maria Vittoria Hospital (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Principal Investigator, Enrico Cecchi, Principal Investigator, Maria Vittoria Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol RF-2013-020358691
Record Dates: First submitted 2017-12-22; First posted 2018-01-26 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Endocarditis
Keywords: Adult; Endocarditis/surgery; Embolism/prevention & control; Cardiovascular Diseases; Costs and Cost Analysis; Quality of life
MeSH Terms: conditions — Endocarditis; Embolism; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Partially Randomized Preference Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early surgery (Experimental): Surgery within 72 hours from endocarditis diagnosis
  Interventions: Procedure: Early surgery
- Conventional therapy (Active Comparator): Medical treatment and a possible delayed surgical intervention according to the current guidelines
  Interventions: Procedure: Conventional therapy

INTERVENTIONS:
Procedure: Early surgery — Surgery within 72 hours from endocarditis diagnosis
  Arms: Early surgery
Procedure: Conventional therapy — Delayed surgical intervention or medical treatment according to the current guidelines
  Arms: Conventional therapy

SUMMARY:
The purpose of the EARLY study is to evaluate the efficacy and effectiveness of early surgery in patients with Infective Endocarditis (IE).

DETAILED DESCRIPTION:
Infective endocarditis (IE) is a relatively rare disease and has a high in-hospital mortality (15-30%) and morbidity due to complications like embolic events, especially in the central nervous system, and heart failure. International guidelines give indications on the optimal timing for surgery, and they strongly recommend early surgery for patients in the active phase of IE with acute cardiac complications (e.g., acute heart failure, uncontrolled infection, and persistent large vegetations after an embolic event). However, at present there is no clear evidence supporting the effectiveness of early surgery or indicating the best time to perform surgery, especially in patients without such conditions. Primary objective of the study is to evaluate whether, in patients with IE and no emergency surgery indication, an early surgical strategy (performed within 72 hours from IE diagnosis) is more effective than conventional therapy in terms of 1-year stroke-free survival. Secondary objectives are: overall survival, risk of embolic, risk of strokes, event-free survival, IE relapse, heart failure, length of hospital stay, hospital re-admission and hospitalization days, strategy compliance, quality of life and health care costs.

This study design consist of a two-arm, open-label, multicenter randomized controlled trial, but patients who decline to be randomized and prefer a certain therapy strategy will be treated according to best practice and included into a prospective observational study after given informed consent. This parallel constructed observational study will be performed with a maximum of consistency to treatment and observation compared to the Randomized clinical trial (RCT). Patients who agree to the randomized trial will be stratified according to centre and clinical features (prosthetic valve,vegetations, valve regurgitation) and randomized with a 1: 1 ratio to 2 different strategies.

According to O'Brien and Fleming group sequential design with a maximum of two stages and a drop-out rate of 10%, a total of 400 randomized patients (200 per group) are required to detect an increase in the stroke-free survival from 82% to 89.5% (corresponding to an Hazard Ratio=0.56) considering a significance level of 5% and a power of 80% and expecting a risk for mortality or stroke at one year with standard treatment equal to 0.18.

EARLY study may help to demonstrate early surgery impact on the contemporary management of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Left-sided Infective Endocarditis (IE) according to modified Duke criteria, fulfilling at least one of the following features:

   * IE on native or prosthetic valve with severe mitral or aortic valve regurgitation, without heart failure;
   * IE on native or prosthetic valve, during the first week of antibiotic therapy, have very large (15-30 mm) or large (>10mm), mobile isolated vegetations due to Staphylococcus aureus, Streptococcus bovis, HACEK or Abiotrophia, without any other indication for surgery;
   * IE on native or prosthetic valve with severe valve regurgitation without heart failure and with large vegetations (> 10 mm) and Euroscore I 5-19;
   * IE on native or prosthetic valve with moderate o moderate-severe valve regurgitation with large vegetations (> 10 mm)
   * IE on prosthetic valve due to Staphylococcus aureus or gram negative non HACEK microorganisms.
2. Compliance to study treatments
3. Euroscore I <20
4. Informed consent signature

Exclusion Criteria:

1. Patients with right-side IE and IE on a cardiac device
2. Patients with IE and:

   * heart failure , refractory pulmonary oedema, cardiogenic shock or untreatable heart failure
   * fistula involving cardiac chambers or pericardium
   * persistent heart failure or unstable echocardiographic signs or poor haemodynamic tolerance
   * uncontrolled local infection (abscess, pseudoaneurism, fistula, increase in size vegetations)
   * fever and positive blood cultures lasting >7 days
   * fungal IE or other multi-resistant microorganisms
   * large vegetations (> 10 mm) after embolic event
   * large vegetations (> 10 mm) and other predictors of complicated course (heart failure, abscess)
   * vegetations >30 mm

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Stroke-free survival | 12 months
  Time from randomization until the first occurrence of stroke or death. Stroke is defined as a focal neurologic deficit, lasting at least 24 hours and is categorized as ischemic, hemorrhagic or of uncertain type.

SECONDARY OUTCOMES:
Overall survival | 12 months
  Time from randomization until death from any cause
In-hospital mortality | During follow-up, until discharge from hospital, up to 1 year from randomization date
  Proportion of death during the hospitalization of IE diagnosis
Embolic event during the hospitalization of IE diagnosis | During follow-up, until discharge from hospital, up to 1 year from randomization date
  Proportion of patients with clinical and instrumental diagnosis of embolic events after IE diagnosis during the same hospitalization
Stroke during the hospitalization of IE diagnosis | During follow-up, until discharge from hospital, up to 1 year from randomization date
  Proportion of patients with clinical and instrumental diagnosis of stroke during the hospitalization of IE diagnosis. Stroke is defined as a focal neurologic deficit, lasting at least 24 hours and is categorized as ischemic, hemorrhagic or of uncertain type.
Heart failure during the hospitalization of IE diagnosis | During follow-up, until discharge from hospital, up to 1 year from randomization date
  Proportion of patients with diagnosis of Heart failure during the hospitalization of IE diagnosis.
Cumulative incidence of stroke | 12 months
  Probability that a patient will have a stroke at 12 months from randomization assuming they do not die from some other cause.
Cumulative incidence of embolic events | 12 months
  Probability that a patient will have an embolic events at 12 months from randomization assuming they do not die from some other cause.
Cumulative incidence of heart failure | 12 months
  Probability that a patients will have a heart failure at 12 months from randomization assuming they do not die from some other cause.
Cumulative incidence of IE relapse | 12 months
  Probability that a patient will have an IE relapse at 12 months from randomization assuming they do not die from some other cause.
Quality of Life using 36-Item Short Form Survey (SF-36) | 0, 4, 12 months
  SF-36 is a generic 36-item questionnaire measuring health-related quality of life (HRQL) composed by 8 subscales. Participants self-report on items that have between 2-6 choices per item using Likert-type responses. Summations of item scores of the same subscale give the subscale scores. Two composite scores, physical component summary (PCS) and mental component summary (MCS), can be derived by a linear combination of the 8 subscales.
  The PCS is represented by 4 subscales: physical function, role limitations due to physical problems, pain, and general health perception. The MCS is represented by 4 subscales: vitality, social function, role limitations due to emotional problems, and mental health.
  Both subscales and composite scores are transformed into a range from 0 to 100; zero= worst HRQL, 100=best HRQL.
Quality of Life using EuroQol five dimension (EQ-5D). | 0, 4, 12 months
  Quality of life will be evaluated using EuroQol five dimension (EQ-5D), a patient-completed, multidimensional measure of health related quality of life. The instrument is applicable to a wide range of health conditions and treatments and results in a single index score. The EQ-5D descriptive health profile comprises five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each dimension comprises three levels (no problems, some/moderate problems, extreme problems). A unique EQ-5D health state is defined by combining one level from each of the five dimensions. EQ-5D index values range from -0.38 to 1.00 (Italian utility weights). Higher EQ-5D Index scores represent better health status.
1-year event-free survival | 12 months
  Time from randomization until the first occurrence of one of the following event: , embolic event, IE relapse and heart failure or death.
Cost-effectiveness | 12 months
  Incremental cost-effectiveness ratio calculated as the ratio between difference in costs and difference in Quality Adjusted Life Years, from EQ-5D (QALYs) among the treatment groups, during the first year after randomization
Length of hospitalization | During follow-up, until discharge from hospital, up to 1 year from randomization date
  Number of days from the date of the randomization and the discharge date
Number of hospital readmission for length .of stay within 1 year for any cause | 12 months
  Number of days of hospitalization for any cause from the the date of discharge
Feasibility of early surgery | During follow-up, until discharge from hospital, up to 1 year from randomization date
  Ratio between the number of patients randomized to early surgery arm and operated within 72 hours and the number of patients randomized to early surgery arm

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Cecchi, MD, Principal Investigator — Maria Vittoria Hospital
Locations (1):
- SC Cardiochirurgia U - AOU Città della Salute e della Scienza di Torino - PO Molinette, Torino, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A web application to collect data for experimental studies — https://www.epiclin.it/early